CLINICAL TRIAL: NCT04361422
Title: Evaluation of the Safety and Efficacy of Isotretinoin in Treatment of COVID-19: Clinical Study
Brief Title: Isotretinoin in Treatment of COVID-19
Acronym: Randomized
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Lamia Elgarhy, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9469305c
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: Isotretinoin; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Isotretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Isotretinoin (Active Comparator): 13 cis retinoic acid 0.5 mg/kg/day in 2 divided doses orally for one month
  Interventions: Drug: Isotretinoin Only Product in Oral Dose Form
- Standard COVID-19 therapy (Sham Comparator): Paracetamol 500 mg /6h, Hydroxychloroquine 500 mg/ 12h, Oseltamivir 150 mg /12 h for 5 days, Azithromycin 1 gm first day then 500 mg/day for 1st line or Clarithromycin 500 mg/12 h for 7-14 days, Ascorbic acid 500 mg/12 h and Cyanocobalamin IV once daily plus Lopinavir 400mg/Ritonavir 100 mg caps 2 capsules twice daily in severe cases
  Interventions: Drug: Isotretinoin Only Product in Oral Dose Form
- Standard COVID-19 therapy+ isotretinoin (Active Comparator): Paracetamol 500 mg /6h, Hydroxychloroquine 500 mg/ 12h, Oseltamivir 150 mg /12 h for 5 days, Azithromycin 1 gm first day then 500 mg/day for 1st line or Clarithromycin 500 mg/12 h for 7-14 days, Ascorbic acid 500 mg/12 h and Cyanocobalamin IV once daily plus Lopinavir 400mg/Ritonavir 100 mg caps 2 capsules twice daily in severe cases) plus 13 cis retinoic acid 0.5 mg/kg/day in 2 divided doses orally forone month.
  Interventions: Drug: Isotretinoin Only Product in Oral Dose Form

INTERVENTIONS:
Drug: Isotretinoin Only Product in Oral Dose Form — assess antiviral efficacy, tolerability and safety of oral isotretinoin in the treatment of COVID-19 versus combined oral isotretinoin with standard therapy for COVID-19 versus the standard therapy alone.
  Other Names: standard COVID-19 therapy

SUMMARY:
Contributors:

Lamia Elgarhy, Sabah El-Gaeish 1, Eman Hamed 2 , Wagdy Fathy2 Department of Dermatology, Department of Pharmacology1 , Faculty of Medicine, Tanta University, Department of Chest, Faculty of Medicine, Suez Canal University2.

Abstract:

The COVID-19 pandemic caused by SARS-COV-2 has infected over 2,000,000 people causing over 150,000 deaths. A key host cellular protein required for the virus entry is angiotensin-converting enzyme 2 (ACE2) whose expression has been demonstrated in many tissues including alveolar epithelial type II cells in lungs, oral mucosa and intestine, heart, kidney, endothelium and skin. ACE2-expressing cells can act as home cells and are prone to SARS-CoV-2 infection as ACE2 receptor facilitates cellular viral entry and replication. (1) Fang et al. has suggested that patients with hypertension and diabetes mellitus may be at higher risk of SARS-CoV-2 infection, as these patients are often treated with ACE inhibitors (ACEIs) or angiotensin II type-I receptor blockers (ARBs), which have been previously suggested to increase ACE2 expression. (2) In another study by Sinha et al who analyzed a publicly available Connectivity Map (CMAP) dataset of pre/post transcriptomic profiles for drug treatment in cell lines for over 20,000 small molecules, isotretinoin was the strongest down-regulator of ACE 2 receptors. On the other hand, they found 6 drugs in CMAP that are currently being investigated in clinical trials for treating COVID-19 (chloroquine, thalidomide, methylprednisolone, losartan, lopinavir and ritonavir, from clinicaltrials.gov), none of which was found to significantly alter ACE2 expression (P>0.1) (3) Moreover, Wu et al, demonstrated that isotretinoin is a Potential papain like protease (PLpro) inhibitors which is a protein encoded by SARS-CoV-2 genes and considered one of the proteins that should be targeted in COVID-19 treatment by performing target-based virtual ligand screening. (4) In addition, isotretinoin was reported to increase CD4 counts and markedly decrease viremia in HIV positive patients suffering from acne vulgaris. (5) Currently, a study is running to evaluate the effect of isotretinoin on immune activation among HIV-1 infected subjects with incomplete CD4+ T cell recovery. (6) From this point, we can suggest that patient taking isotretinoin therapy may be immune against SARS-COV-2 and it can also have a therapeutic effect by prevention of further progression of the virus. Several potential mechanisms of action of Chloroquine/Hydroxychloroquine against SARS-CoV-2 have been postulated and they are actually used in treatment regimens for COVID-19.(7) It was reported that chloroquine increase the blood level of isotretinoin, so lower doses is required when combined. We assume to test the efficacy of isotretinoin in treatment of COVID-19 versus combined therapy with the standard treatment of COVID-19.

DETAILED DESCRIPTION:
The study is a randomized interventional comparative Phase III trial. The duration of the trial for each subject is expected to be 3 months. The duration for each individual subject includes one-month study treatment and 3 months follow-up time. Recruitment of subjects will start in April 2020.

150 adult male and female patients with positive COVID-19 diagnosis and fulfilling the below outlined inclusion criteria will be enrolled into the study. Trial population will consist of both genders.

Name of tested drug: Isotretinoin. All consenting adult patients having confirmed COVID-19 will be recruited and randomly and blindly allocated in a 1:1:1 ratio to the following arms:

Group (1): 50 patients will receive isotretinoin 0.5 mg/kg/day for one month or until viral clearance.

Group (2): 50 patients will receive standard therapy for COVID-19 (Paracetamol 500 mg /6h, Hydroxychloroquine 500 mg/ 12h, Oseltamivir 150 mg /12 h for 5 days, Azithromycin 1 gm first day then 500 mg/day for 1st line or Clarithromycin 500 mg/12 h for 7-14 days, Ascorbic acid 500 mg/12 h and Cyanocobalamin IV once daily plus Lopinavir 400mg/Ritonavir 100 mg caps 2 capsules twice daily in severe cases).

Group (3): 50 patients will receive standard therapy for COVID-19 + isotretinoin 0.25 mg/kg/day for one month or until viral clearance.

Inclusion Criteria:

* Clinical and laboratory diagnosis of COVID-19.
* Age range 18-40

Exclusion Criteria:

• Have the following conditions:

1. Hypercholesterolemia
2. Hypertriglyceridemia
3. Liver disease
4. Renal disease
5. Sjögren syndrome
6. Pregnancy
7. Lactation
8. Depressive disorder
9. Contraindications for hormonal contraception or intrauterine device.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of COVID-19.
* Age range 18-40

Exclusion Criteria:

1. Hypercholesterolemia
2. Hypertriglyceridemia
3. Liver disease
4. Renal disease
5. Sjögren syndrome
6. Pregnancy
7. Lactation
8. Depressive disorder
9. Contraindications for hormonal contraception or intrauterine device.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical clearance | 14-30 day
  1. Difference in time to resolution of clinical signs and symptoms of COVID-19 treated with isotretinoin, standard therapy or combined therapy as assessed by daily assessment

OTHER OUTCOMES:
Laboratory clearance | 14-30 day
  1. Proportion of patients with negative COVID-19 PCR test at day 30 in per protocol population as per throat swab
  2. Change in COVID-19 virus load from baseline to day 30

IPD SHARING:
Plan to Share IPD: No